CLINICAL TRIAL: NCT03353558
Title: OBJECTIVE AND SUBJECTIVE ASSESSMENT OF SLEEP QUALITY IN PATIENTS WITH CHRONIC MYELOGENOUS LEUKEMIA
Brief Title: Sleep Assessment in CML
Acronym: CML-SLEEP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: The Max Stern Academic College Of Emek Yezreel (Other)
Responsible Party: Principal Investigator, Ariel Aviv, Head of hematology, HaEmek Medical Center, Israel
Other Study IDs: EMC 141-17
Record Dates: First submitted 2017-11-16; First posted 2017-11-27 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Sleep Disorder; Chronic Myeloid Leukemia
MeSH Terms: conditions — Sleep Wake Disorders; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Study Group (CML group): This group will be CML patients. In this group each participant will be asked to wear a watch "Actigraph" for one week.
  He will be asked to fill the appropriate questionnaires, and a daily sleep diary.
  Interventions: Device: Actigraph
- Control Group: The control group will be non-CML patients, also without any known malignancy or known sleep disturbances.
  They will be asked to wear the watch "Actigraph" for one week, and to fill the appropriate questionnaires and a daily sleep diary.
  Interventions: Device: Actigraph

INTERVENTIONS:
Device: Actigraph — The watch will measure sleep parameters like quality of sleep, time to fall asleep, number of awakenings during night, length of deep sleep.
  Other Names: Actiwatch (different name for the same device)

SUMMARY:
Patients with CML report on fatigue, and many of them report on sleep disturbances. The investigators wish to objectively assess the patient's sleep using a sleep "wrist watch" (Actigraph) , and correlate data with their perception of sleep quality. A matched participants group will serve as control. the Control group is defined as participants not having CML or any other malignancy and without any known sleep disturbances.

DETAILED DESCRIPTION:
The investigators will contact the CML patients cohort (about 50) and ask them to join the study. Those consenting will be briefed on the use of an Actigraph wrist device, which the patients should wear for a week. In addition, patients will fill quality of life, depression and anxiety questionnaires.

During the assessment week they will be asked to fill in a short "sleep diary" to be correlated with the objective Actigraph results.

The investigators will analyze objective data and compare to the subjective report of patient's sleep and compare these results with a matched cohort of the control participants. The investigators will analyze the quality of life, anxiety and depression scores also.

The main objective of the study is to try and find a correlation between CML and sleep disturbances, several previous studies found sleep disturbances in reported questionnaires, but the sleep parameters were never studied objectively. Also most of the studies concentrated on the fatigue as the main symptom, in our study the investigators will focus on sleep quality and quantity as a primary symptom.

The quality of life questionnaire will be WHOQOL-BREF questionnaire. The anxiety questionnaire will be Hamilton Anxiety Rating Scale. The depression questionnaire will be Beck Depression Inventory.

The sleep watch that will be used is called Actigraph/Actiwatch and it is FDA approved device, this device will help the investigators assess and observe the objective sleep parameters like length of sleep, time to fall asleep, number of awakenings at night.

There will be no intervention in the study, the results will not alter the treatment the patients receive. But if some patients will be found to have a severe depression or anxiety they will be referred to psychiatric consult.

the study will be with the collaboration of Professor Iris Haymov, sleep researcher from the Max Stern Academic College of Emek Yezreel.

ELIGIBILITY:
Inclusion Criteria:

* CML patients
* Without known sleep disturbances that are not related to the disease

Exclusion Criteria:

* Malignancy other than CML
* Known sleep disturbances
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CML patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of subjective and objective sleep disturbances among patients with CML | 1 week of sleep parameters measuring
  The prevalence will be compared to the Control group in the study and to the prevalnce of sleep disturbances reported in other studies.

SECONDARY OUTCOMES:
Comparison between the subjective sleep disturbances reported and the objective sleep disturbances measured in the CML patients group. | 1 week
  The investigators will correlate between the subjective and the objective results. the investigators will seek correlation between the anxiety, quality of life and depression questionnaires and the subjective reports of sleep disturbances and whether these reports supported objectively or not
Correlation of objective sleep disturbances with the CML patients characteristics. | 1 week
  The characteristics that will be used will be: the duration of the disease, the clinical response to therapy, the type of therapy that the patients receive.

CONTACTS AND LOCATIONS:
Overall Officials: Aviv A Ariel, Doctor, Principal Investigator — Head of hematology department

IPD SHARING:
Plan to Share IPD: Yes
All date can be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available as from December 2018. The data will be available all the time.
Access Criteria: Anyone can access